CLINICAL TRIAL: NCT06711627
Title: Arkansas Community Engagement Alliance: Delivering Arkansas Perinatal Outcomes for Minority and Rural Women Through Innovative System Improvement to Create Equity
Brief Title: Food Provision in Prenatal Care
Acronym: FPPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 297889
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy Complications; Excessive Gestational Weight Gain
MeSH Terms: conditions — Pregnancy Complications | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SoC) (Active Comparator): The SoC arm includes implementing the standard clinical protocol for nutritional and gestational weight gain counseling recommended for all pregnant women. Additionally, participants in the SoC arm will receive $500 after delivery to be used for baby items.
  Interventions: Behavioral: Standard of Care (SoC)
- Food Provision (Experimental): The Food Provision arm includes the same nutritional and gestational weight gain counseling provided as standard of care. In addition, participants in the Food Provision arm will be provided with a total of $1000 during their pregnancy to be used specifically for the purchase of healthy foods.
  Interventions: Behavioral: Food Provision

INTERVENTIONS:
Behavioral: Standard of Care (SoC) — Standard recommended nutrition and gestational weight gain counseling.
  Arms: Standard of Care (SoC)
Behavioral: Food Provision — Standard recommended nutrition and gestational weight gain counseling plus food provision.
  Arms: Food Provision

SUMMARY:
The overarching research question is: "Does the provision of healthy food during pregnancy reduce the proportion of women who experience excessive gestational weight gain compared with standard of care (SoC)?" To answer this question, the investigators will conduct a randomized controlled trial with 400 pregnant women. Participants will be randomized 1:1 to either the Food Provision arm or the SoC arm, with approximately 200 participants per arm. Participants randomized to the SoC arm will receive the standard clinical protocol for nutritional and gestational weight gain counseling recommended for all pregnant women, as well as $500 after delivery to be used specifically for baby items.Those randomized to the Food Provision arm will be provided the same nutritional and gestational weight gain counseling, as well as a total of $1000 during pregnancy to be used specifically for the purchase of healthy foods recommended in the nutritional counseling. Data for the primary outcome will be collected from birth records and from surveys conducted at baseline (pre-intervention), midpoint (between 24-36 weeks gestation), and post-intervention (~8 weeks post-partum).

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-44 years
* <= 22 weeks Pregnant
* Speak English, Spanish, or Marshallese
* Valid email address
* Resides in and plans to give birth in the state of Arkansas

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Excessive Gestational Weight Gain (EGWG) | Baseline to Post-partum (approx. 40 weeks)
  Pre-pregnancy weight and weight immediately prior to birth will be used to calculate total weight gain, adjusting for pre-pregnancy body mass index and weeks of gestation. Individuals whose total weight gain exceeds established guidelines will be determined to have EGWG.

CONTACTS AND LOCATIONS:
Locations (1):
- UAMS Institute for Community Health Innovation, Springdale, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No